CLINICAL TRIAL: NCT00005143
Title: Stanford Five-City Multifactor Risk Reduction Study
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1014; R01HL021906 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Atherosclerosis; Coronary Disease; Cerebrovascular Accident; Myocardial Infarction; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Atherosclerosis; Coronary Disease; Stroke; Myocardial Infarction; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To conduct a large-scale demonstration and education project designed to evaluate the feasibility and effectiveness of long-term community health education directed toward lowering cardiovascular disease risk, morbidity, and mortality. Targeted risk factors included general lifestyle, smoking, blood pressure, nutrition and weight, and exercise. The program was evaluated by biennial cross-sectional independent surveys, longitudinal studies, and morbidity and mortality surveillance.

DETAILED DESCRIPTION:
BACKGROUND:

The last fifty years of research into cardiovascular diseases have shown strong associations between individual risk factor levels and disease rates within and among many cultures. The potential for medical treatment of cardiovascular disease is limited by the insidious development of atherosclerosis and hypertension, the high immediate mortality of coronary disease and stroke, and the inadequacy of treatment for the advanced stages of cardiovascular disease. All of these factors, coupled with the predictable safety and general feasibility of individual risk factor reduction, provided the stimulus for developing community-wide strategies for the prevention of cardiovascular disease.

The Stanford Three Community Study, conducted between 1972 and 1975, and the Five City Project (FCP) were designed to test the feasibility and effectiveness of such community-wide preventive approaches. Both the Three Community Study and the Five City Project have shown that risk factors can be reduced on a community-wide level, particularly smoking rates and blood pressure levels. These studies were congruent with other contemporary studies, such as the Belgium Heart Disease Prevention Project and the North Karelia Project.

Despite these successes, however, there were additional questions. Would the reduction in risk be translated into a reduction in morbidity and mortality? The North Karelia Project was apparently associated with a fall in mortality as was the Belgium Heart Disease Prevention Program. However, the U.K. Heart Disease Prevention Project was not effective nor was the Multiple Risk Factor Intervention Trial in reducing mortality. It is an appropriate responsibility of the scientific community to inform the general public of the implications of this research and to give advice on the prudent preventive measures.

DESIGN NARRATIVE:

The study had a quasi-experimental design with two California cities, Salinas and Monterey, selected as intervention cities and three similar cities, San Luis Obispo, Modesto, and Santa Monica as control cities. The selection of cities was subject to several criteria including: location in Northern California; population exceeding 30,000 with a total of all five cities exceeding 300,000 to provide sufficient statistical power; ethnic, socioeconomic and demographic similarity; independence from other cities; no shared newspaper or electronic media between treatment and control cities and shared media markets between treatment cities; and independence of the two treatment cities. The education program began in 1980 after the completion of a baseline population survey and continued for eight years. Education methods included the use of television and radio, newspapers, books, pamphlets, and community programs developed through health departments, schools, voluntary organizations, hospitals and non-profit health service agencies.

The effectiveness of the program was evaluated by population surveys in Monterey, Salinas, Modesto, and San Luis Obispo but not Santa Monica and by a morbidity and mortality surveillance system. In the initial year of the survey in 1979-1980, approximately 600 people in each community visited the survey center. This comprised the first independent sample of the community. After an average of 15 months, these same individuals returned to the survey center for a follow-up evaluation. This cohort sample has been studied every other year for five surveys to determine the process of change in cardiovascular risk and related behaviors over time. Five randomly-selected independent samples have been surveyed to study cross-sections of the community over time. Questionnaires and dietary measures were the chief sources of data on health-related behaviors. The questionnaire contained components on: demographic measures; attitude and opinion measures; health knowledge assessment related to prevention of heart disease and stroke; stress behavior; diet, nutrition, and weight behavior; smoking behavior; physical activity behavior; communication media use; and medical history including medication use. A random 40 percent of the initial sample completed a 24-hour dietary recall which was re-administered in the fourth cohort survey and was also administered to a 50 percent random sample of the fourth independent survey. Biological measurements consisted of height and weight, blood pressure, resting heart rate, plasma thiocyanate, total cholesterol, triglycerides and cholesterol content of lipoprotein subfractions, expired air carbon dioxide, urinary sodium, potassium and creatinine, and an exercise test. Data were also collected on plasma apolipoprotein A-1 and B and on high density lipoprotein subfractions 2 and 3. A comprehensive dietary assessment was also conducted.

Community surveillance was conducted to allow the calculation of comparable, city-specific rates for total mortality, cardiovascular mortality, fatal myocardial infarction, nonfatal myocardial infarction, fatal and nonfatal stroke. Development of the community surveillance system was done in close collaboration with the Minnesota Heart Health Project and the Pawtucket Heart Health Project to insure comparability. Only those cardiovascular disease events which always resulted in hospitalization were monitored and included myocardial infarction and stroke. Fatal cases were identified from county death certificate files. Both fatal and nonfatal hospitalized events were investigated by abstracting the medical records onto a set of standard forms. All non-hospitalized deaths were investigated by contacting the decedent's family for medical history and circumstances of death and by contacting the decedent's physician for medical information. Data were monitored on the severity of coronary events and on the quality of care. An Acute Coronary Care form was designed in cooperation with the Minnesota surveillance project and with the MONICA project. The form was field tested in September 1985 and was implemented retroactively on 1980 and 1981 cases.

The study was renewed in 1992 to 1) extend morbidity and mortality surveillance by three years (to June 1994 for events through December 1992); 2) to extend analysis and publication of Five City Project (FCP) results and methods; and 3) to provide a small amount of incremental support to enable use of frozen plasma samples from earlier FCP population surveys to conduct a nested case-control study of the association of HDL subfractions and apolipoproteins with fatal and non-fatal cardiovascular disease. Extension of surveillance data collection was needed to insure the detection of any impact on morbidity and mortality of the significant risk factor changes that occurred in the treatment cities, compared to control cities, by 1986. The nested case-control study involved matching the survey and surveillance data sets to identify persons with documented events who participated in one of the five population surveys, identifying and contacting potential controls to be certain that they were free of CVD, and analysis of plasma samples frozen at -80 degrees centigrade for apolipoproteins A-I and B and HDL2,3 subfractions. This allowed multifactor assessment of the association between those factors and CVD in persons for whom many other variables were known.

ELIGIBILITY:
No eligibility criteria

Ages: 0 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2504 (Actual)
Dates: Start 1978-07 (Actual); Primary Completion 1994-07 (Actual); Study Completion 1994-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John W Farquhar, Principal Investigator — Stanford University

REFERENCES:
- [Background] Farquhar JW, Fortmann SP, Maccoby N, Wood PD, Haskell WL, et al: The Stanford Five City Project: An Overview. In: Matarazzo JD, Miller NE, Weiss SM, Herd JA & Weiss SM (Eds), Behavioral Health: A Handbook of Health Enhancement and Disease Prevention. John Wiley & Sons, Inc., Silver Spring, MD, 1154-1165, 1984
- [Background] Fortmann SP, Rogers T, Vranizan K, Haskell WL, Solomon DS, Farquhar JW. Indirect measures of cigarette use: expired-air carbon monoxide versus plasma thiocyanate. Prev Med. 1984 Jan;13(1):127-35. doi: 10.1016/0091-7435(84)90045-8. PMID 6609353
- [Background] Solomon DS, Maccoby N: Communication as a Model for Health Enhancement. In: Matarazzo JD, Miller NE, Weiss SM, Herd JA and Weiss SM (Eds), Behavioral Health: A Handbook of Health Enhancement and Disease Prevention. Silver Spring, MD: John Wiley, Chapter 13, pp. 209-221, 1984
- [Background] Sallis JF, Haskell WL, Wood PD, Fortmann SP, Rogers T, Blair SN, Paffenbarger RS Jr. Physical activity assessment methodology in the Five-City Project. Am J Epidemiol. 1985 Jan;121(1):91-106. doi: 10.1093/oxfordjournals.aje.a113987. PMID 3964995
- [Background] Sallis JF, Flora JA, Fortmann SP, Taylor CB, Maccoby N. Mediated smoking cessation programs in the Stanford Five-City Project. Addict Behav. 1985;10(4):441-3. doi: 10.1016/0306-4603(85)90043-7. PMID 4091078
- [Background] Farquhar JW, Fortmann SP, Maccoby N, Haskell WL, Williams PT, Flora JA, Taylor CB, Brown BW Jr, Solomon DS, Hulley SB. The Stanford Five-City Project: design and methods. Am J Epidemiol. 1985 Aug;122(2):323-34. doi: 10.1093/oxfordjournals.aje.a114104. PMID 4014215
- [Background] Blair SN, Haskell WL, Ho P, Paffenbarger RS Jr, Vranizan KM, Farquhar JW, Wood PD. Assessment of habitual physical activity by a seven-day recall in a community survey and controlled experiments. Am J Epidemiol. 1985 Nov;122(5):794-804. doi: 10.1093/oxfordjournals.aje.a114163. PMID 3876763
- [Background] Fortmann SP, Sallis JF, Magnus PM, Farquhar JW. Attitudes and practices of physicians regarding hypertension and smoking: The Stanford Five City Project. Prev Med. 1985 Jan;14(1):70-80. doi: 10.1016/0091-7435(85)90022-2. PMID 4034516
- [Background] Farquhar JW, Maccoby N, Wood PD: Education and Communication Studies. In: Holland WW, Detels R & Knox G (Eds). Oxford Textbook of Public Health0, Vol. 3. Oxford, London: Oxford University Press, pp. 207-221, 1985
- [Background] Jacob RG, Fortmann SP, Kraemer HC, Farquhar JW, Agras WS. Combining behavioral treatments to reduce blood pressure. A controlled outcome study. Behav Modif. 1985 Jan;9(1):32-53. doi: 10.1177/01454455850091003. No abstract available. PMID 3977813
- [Background] Sallis JF, Haskell WL, Wood PD, Fortmann SP, Vranizan KM. Vigorous physical activity and cardiovascular risk factors in young adults. J Chronic Dis. 1986;39(2):115-20. doi: 10.1016/0021-9681(86)90067-6. PMID 3484748
- [Background] Fortmann SP, Haskell WL, Williams PT, Varady AN, Hulley SB, Farquhar JW. Community surveillance of cardiovascular diseases in the Stanford Five-City Project. Methods and initial experience. Am J Epidemiol. 1986 Apr;123(4):656-69. doi: 10.1093/oxfordjournals.aje.a114285. PMID 3953544
- [Background] Fortmann SP, Haskell WL, Williams PT. Changes in plasma high density lipoprotein cholesterol after changes in cigarette use. Am J Epidemiol. 1986 Oct;124(4):706-10. doi: 10.1093/oxfordjournals.aje.a114445. No abstract available. PMID 3752064
- [Background] Sallis JF, Hill RD, Killen JD, Telch MJ, Flora JA, Girard J, Taylor CB, Fortmann SP. Efficacy of self-help behavior modification materials in smoking cessation. Am J Prev Med. 1986 Nov-Dec;2(6):342-4. PMID 3453200
- [Background] Sallis JF, Haskell WL, Fortmann SP, Wood PD, Vranizan KM. Moderate-intensity physical activity and cardiovascular risk factors: the Stanford Five-City Project. Prev Med. 1986 Nov;15(6):561-8. doi: 10.1016/0091-7435(86)90061-7. PMID 3797388
- [Background] Sallis JF, Hill RD, Fortmann SP, Flora JA. Health behavior change at the worksite: cardiovascular risk reduction. Prog Behav Modif. 1986;20:161-97. doi: 10.1016/b978-0-12-535620-6.50009-3. No abstract available. PMID 3517827
- [Background] Sallis JF, Haskell WL, Fortmann SP, Vranizan KM, Taylor CB, Solomon DS. Predictors of adoption and maintenance of physical activity in a community sample. Prev Med. 1986 Jul;15(4):331-41. doi: 10.1016/0091-7435(86)90001-0. PMID 3763558
- [Background] Chafee SH, Roser C: Involvement and the Consistency of Knowledge, Attitudes, and Behaviors. Commun Res, 13:373-399, 1986
- [Background] King AC, Flora JA, Fortmann SP, Taylor CB. Smokers' challenge: immediate and long-term findings of a community smoking cessation contest. Am J Public Health. 1987 Oct;77(10):1340-1. doi: 10.2105/ajph.77.10.1340. PMID 3631371
- [Background] Tuomilehto J, Kuulasmaa K, Torppa J. WHO MONICA Project: geographic variation in mortality from cardiovascular diseases. Baseline data on selected population characteristics and cardiovascular mortality. World Health Stat Q. 1987;40(2):171-84. No abstract available. English, French. PMID 3617777
- [Background] Maron DJ, Fortmann SP. Nicotine yield and measures of cigarette smoke exposure in a large population: are lower-yield cigarettes safer? Am J Public Health. 1987 May;77(5):546-9. doi: 10.2105/ajph.77.5.546. PMID 3565645
- [Background] Altman DG, Flora JA, Fortmann SP, Farquhar JW. The cost-effectiveness of three smoking cessation programs. Am J Public Health. 1987 Feb;77(2):162-5. doi: 10.2105/ajph.77.2.162. PMID 3099586
- [Background] Williams PT, Karlin S, Farquhar JW. Permutation analyses of familial association arrays for lipoprotein concentrations in families of the Stanford Five City Project. Am J Epidemiol. 1987 Dec;126(6):1126-40. doi: 10.1093/oxfordjournals.aje.a114751. PMID 3687922
- [Background] King AC, Saylor KE, Foster S, Killen JD, Telch MJ, Farquhar JW, Flora JA. Promoting dietary change in adolescents: a school-based approach for modifying and maintaining healthful behavior. Am J Prev Med. 1988 Mar-Apr;4(2):68-74. PMID 3395493
- [Background] Flora JA, Farquhar JW. Methods of message design: experiences from the Stanford Five City Project. Scand J Prim Health Care Suppl. 1988;1:39-47. PMID 3227201
- [Background] Farquhar JW, Fortmann SP, Flora JA, Taylor CB, Haskell WL, Williams PT, Maccoby N, Wood PD. Effects of communitywide education on cardiovascular disease risk factors. The Stanford Five-City Project. JAMA. 1990 Jul 18;264(3):359-65. PMID 2362332
- [Background] Fortmann SP, Winkleby MA, Flora JA, Haskell WL, Taylor CB. Effect of long-term community health education on blood pressure and hypertension control. The Stanford Five-City Project. Am J Epidemiol. 1990 Oct;132(4):629-46. doi: 10.1093/oxfordjournals.aje.a115705. PMID 2403104
- [Background] Albright CL, Flora JA, Fortmann SP. Restaurant menu labeling: impact of nutrition information on entree sales and patron attitudes. Health Educ Q. 1990 Summer;17(2):157-67. doi: 10.1177/109019819001700203. PMID 2347693
- [Background] Winkleby MA, Fortmann SP, Barrett DC. Social class disparities in risk factors for disease: eight-year prevalence patterns by level of education. Prev Med. 1990 Jan;19(1):1-12. doi: 10.1016/0091-7435(90)90001-z. PMID 2320553
- [Background] Frank E, Winkleby MA, Fortmann SP, Rockhill B, Farquhar JW. Improved cholesterol-related knowledge and behavior and plasma cholesterol levels in adults during the 1980s. JAMA. 1992 Sep 23-30;268(12):1566-72. PMID 1518111
- [Background] Taylor CB, Fortmann SP, Flora J, Kayman S, Barrett DC, Jatulis D, Farquhar JW. Effect of long-term community health education on body mass index. The Stanford Five-City Project. Am J Epidemiol. 1991 Aug 1;134(3):235-49. doi: 10.1093/oxfordjournals.aje.a116077. PMID 1877583
- [Background] Farquhar JW. The Stanford Cardiovascular Disease Prevention Programs. Ann N Y Acad Sci. 1991;623:327-31. doi: 10.1111/j.1749-6632.1991.tb43742.x. No abstract available. PMID 2042841
- [Background] Winkleby MA, Fortmann SP, Rockhill B. Trends in cardiovascular disease risk factors by educational level: the Stanford Five-City Project. Prev Med. 1992 Sep;21(5):592-601. doi: 10.1016/0091-7435(92)90067-r. PMID 1438109
- [Background] Hyman DJ, Barrett DC, Fortmann SP. Effect of minor illness on serum cholesterol level. Am J Prev Med. 1992 Mar-Apr;8(2):100-3. PMID 1599716
- [Background] Winkleby MA, Jatulis DE, Frank E, Fortmann SP. Socioeconomic status and health: how education, income, and occupation contribute to risk factors for cardiovascular disease. Am J Public Health. 1992 Jun;82(6):816-20. doi: 10.2105/ajph.82.6.816. PMID 1585961
- [Background] Jackson C, Jatulis DE, Fortmann SP. The Behavioral Risk Factor Survey and the Stanford Five-City Project Survey: a comparison of cardiovascular risk behavior estimates. Am J Public Health. 1992 Mar;82(3):412-6. doi: 10.2105/ajph.82.3.412. PMID 1536358
- [Background] Jackson C, Winkleby MA, Flora JA, Fortmann SP. Use of educational resources for cardiovascular risk reduction in the Stanford Five-City Project. Am J Prev Med. 1991 Mar-Apr;7(2):82-8. PMID 1910892
- [Background] Williams JE, Flora JA. Health behavior segmentation and campaign planning to reduce cardiovascular disease risk among Hispanics. Health Educ Q. 1995 Feb;22(1):36-48. doi: 10.1177/109019819502200105. PMID 7721600
- [Background] Taylor CB, Jatulis DE, Winkleby MA, Rockhill BJ, Kraemer HC. Effects of life-style on body mass index change. Epidemiology. 1994 Nov;5(6):599-603. doi: 10.1097/00001648-199411000-00007. PMID 7841241
- [Background] Davis SK, Winkleby MA, Farquhar JW. Increasing disparity in knowledge of cardiovascular disease risk factors and risk-reduction strategies by socioeconomic status: implications for policymakers. Am J Prev Med. 1995 Sep-Oct;11(5):318-23. PMID 8573362
- [Background] Fortmann SP, Flora JA, Winkleby MA, Schooler C, Taylor CB, Farquhar JW. Community intervention trials: reflections on the Stanford Five-City Project Experience. Am J Epidemiol. 1995 Sep 15;142(6):576-86. doi: 10.1093/oxfordjournals.aje.a117678. PMID 7653465
- [Background] Frank E, Winkleby M, Fortmann SP, Rockhill B, Farquhar JW. Improvements in cholesterol-related knowledge and behavior and plasma cholesterol levels in youths during the 1980s. Am J Prev Med. 1993 May-Jun;9(3):168-74. PMID 8347368
- [Background] Frank E, Winkleby M, Fortmann SP, Farquhar JW. Cardiovascular disease risk factors: improvements in knowledge and behavior in the 1980s. Am J Public Health. 1993 Apr;83(4):590-3. doi: 10.2105/ajph.83.4.590. PMID 8460744
- [Background] Winkleby MA, Schooler C, Kraemer HC, Lin J, Fortmann SP. Hispanic versus white smoking patterns by sex and level of education. Am J Epidemiol. 1995 Aug 15;142(4):410-8. doi: 10.1093/oxfordjournals.aje.a117649. PMID 7625406
- [Background] Taylor CB, Jatulis DE, Fortmann SP, Kraemer HC. Weight variability effects: a prospective analysis from the Stanford Five-City Project. Am J Epidemiol. 1995 Mar 1;141(5):461-5. doi: 10.1093/oxfordjournals.aje.a117448. PMID 7879790
- [Background] Winkleby MA, Albright CL, Howard-Pitney B, Lin J, Fortmann SP. Hispanic/white differences in dietary fat intake among low educated adults and children. Prev Med. 1994 Jul;23(4):465-73. doi: 10.1006/pmed.1994.1064. PMID 7971874
- [Background] Young DR, Haskell WL, Jatulis DE, Fortmann SP. Associations between changes in physical activity and risk factors for coronary heart disease in a community-based sample of men and women: the Stanford Five-City Project. Am J Epidemiol. 1993 Aug 15;138(4):205-16. doi: 10.1093/oxfordjournals.aje.a116849. PMID 8356962
- [Background] Winkleby MA, Fortmann SP, Rockhill B. Health-related risk factors in a sample of Hispanics and whites matched on sociodemographic characteristics. The Stanford Five-City Project. Am J Epidemiol. 1993 Jun 15;137(12):1365-75. doi: 10.1093/oxfordjournals.aje.a116646. PMID 8333418
- [Background] Williams EL, Winkleby MA, Fortmann SP. Changes in coronary heart disease risk factors in the 1980s: evidence of a male-female crossover effect with age. Am J Epidemiol. 1993 May 15;137(10):1056-67. doi: 10.1093/oxfordjournals.aje.a116609. PMID 8317435
- [Background] Fortmann SP, Taylor CB, Flora JA, Winkleby MA. Effect of community health education on plasma cholesterol levels and diet: the Stanford Five-City Project. Am J Epidemiol. 1993 May 15;137(10):1039-55. doi: 10.1093/oxfordjournals.aje.a116608. PMID 8317434
- [Background] Fortmann SP, Taylor CB, Flora JA, Jatulis DE. Changes in adult cigarette smoking prevalence after 5 years of community health education: the Stanford Five-City Project. Am J Epidemiol. 1993 Jan 1;137(1):82-96. doi: 10.1093/oxfordjournals.aje.a116605. PMID 8434576
- [Background] Farquhar JW, Fortmann SP, Wood PD, Haskell WL: Community Studies of Cardiovascular Disease Prevention. In: Kaplan NM, Stamler J (Eds). Prevention of Coronary Heart Disease. Philadelphia: W.B. Saunders, 170-181, 1983
- [Background] Fortmann SP, Haskell WL, Vranizan K, Brown BW, Farquhar JW. The association of blood pressure and dietary alcohol: differences by age, sex, and estrogen use. Am J Epidemiol. 1983 Oct;118(4):497-507. doi: 10.1093/oxfordjournals.aje.a113655. PMID 6637977
- [Background] Farquhar JW, Maccoby N, Solomon DS: Community Applications of Behavioral Medicine. In: Gentry WD (Ed), Handbook of Behavioral Medicine, The Guilford Press, NY, 437-478, 1984
- [Background] King AC, Kiernan M, Ahn DK, Wilcox S. The effects of marital transitions on changes in physical activity: results from a 10-year community study. Ann Behav Med. 1998 Spring;20(2):64-9. doi: 10.1007/BF02884450. PMID 9989310
- [Background] Greeno CG, Jackson C, Williams EL, Fortmann SP. The effect of perceived control over eating on the life satisfaction of women and men: results from a community sample. Int J Eat Disord. 1998 Dec;24(4):415-9. doi: 10.1002/(sici)1098-108x(199812)24:43.0.co;2-9. PMID 9813766
- [Background] Davis SK, Ahn DK, Fortmann SP, Farquhar JW. Determinants of cholesterol screening and treatment patterns. Insights for decision-makers. Am J Prev Med. 1998 Oct;15(3):178-86. doi: 10.1016/s0749-3797(98)00047-6. PMID 9791635
- [Background] Ribisl KM, Winkleby MA, Fortmann SP, Flora JA. The interplay of socioeconomic status and ethnicity on Hispanic and white men's cardiovascular disease risk and health communication patterns. Health Educ Res. 1998 Sep;13(3):407-17. doi: 10.1093/her/13.3.407. PMID 10186451
- [Background] Winkleby MA, Feldman HA, Murray DM. Joint analysis of three U.S. community intervention trials for reduction of cardiovascular disease risk. J Clin Epidemiol. 1997 Jun;50(6):645-58. doi: 10.1016/s0895-4356(97)00020-6. PMID 9250263
- [Background] Wild SH, Fortmann SP, Marcovina SM. A prospective case-control study of lipoprotein(a) levels and apo(a) size and risk of coronary heart disease in Stanford Five-City Project participants. Arterioscler Thromb Vasc Biol. 1997 Feb;17(2):239-45. doi: 10.1161/01.atv.17.2.239. PMID 9081676
- [Background] Winkleby MA, Taylor CB, Jatulis D, Fortmann SP. The long-term effects of a cardiovascular disease prevention trial: the Stanford Five-City Project. Am J Public Health. 1996 Dec;86(12):1773-9. doi: 10.2105/ajph.86.12.1773. PMID 9003136
- [Background] Oka RK, Fortmann SP, Varady AN. Differences in treatment of acute myocardial infarction by sex, age, and other factors (the Stanford Five-City Project). Am J Cardiol. 1996 Oct 15;78(8):861-5. doi: 10.1016/s0002-9149(96)00457-2. PMID 8888655
- [Background] Gardner CD, Fortmann SP, Krauss RM. Association of small low-density lipoprotein particles with the incidence of coronary artery disease in men and women. JAMA. 1996 Sep 18;276(11):875-81. PMID 8782636
- [Background] Schooler C, Sundar SS, Flora J. Effects of the Stanford Five-City Project Media Advocacy Program. Health Educ Q. 1996 Aug;23(3):346-64. doi: 10.1177/109019819602300306. PMID 8841819
- [Background] Young DR, Haskell WL, Taylor CB, Fortmann SP. Effect of community health education on physical activity knowledge, attitudes, and behavior. The Stanford Five-City Project. Am J Epidemiol. 1996 Aug 1;144(3):264-74. doi: 10.1093/oxfordjournals.aje.a008921. PMID 8686695
- [Background] Winkleby MA, Gardner CD, Taylor CB. The influence of gender and socioeconomic factors on Hispanic/white differences in body mass index. Prev Med. 1996 Mar-Apr;25(2):203-11. doi: 10.1006/pmed.1996.0047. PMID 8860286
- [Background] Winkleby MA, Kraemer H, Lin J, Jatulis D, Fortmann SP. Sociodemographic influences on Hispanic-white differences in blood pressure. Public Health Rep. 1996;111 Suppl 2(Suppl 2):30-2. PMID 8898768
- [Background] Wild SH, Laws A, Fortmann SP, Varady AN, Byrne CD. Mortality from coronary heart disease and stroke for six ethnic groups in California, 1985 to 1990. Ann Epidemiol. 1995 Nov;5(6):432-9. doi: 10.1016/1047-2797(95)00058-5. PMID 8680605
- [Background] Fortmann SP, Varady AN. Effects of a community-wide health education program on cardiovascular disease morbidity and mortality: the Stanford Five-City Project. Am J Epidemiol. 2000 Aug 15;152(4):316-23. doi: 10.1093/aje/152.4.316. PMID 10968376
- [Background] Gardner CD, Tribble DL, Young DR, Ahn D, Fortmann SP. Associations of HDL, HDL(2), and HDL(3) cholesterol and apolipoproteins A-I and B with lifestyle factors in healthy women and men: the Stanford Five City Project. Prev Med. 2000 Oct;31(4):346-56. doi: 10.1006/pmed.2000.0716. PMID 11006059
- [Background] Gardner CD, Tribble DL, Young DR, Ahn D, Fortmann SP. Population frequency distributions of HDL, HDL(2), and HDL(3) cholesterol and apolipoproteins A-I and B in healthy men and women and associations with age, gender, hormonal status, and sex hormone use: the Stanford Five City Project. Prev Med. 2000 Oct;31(4):335-45. doi: 10.1006/pmed.2000.0715. PMID 11006058
- [Background] Rimal RN. Closing the knowledge-behavior gap in health promotion: the mediating role of self-efficacy. Health Commun. 2000;12(3):219-37. doi: 10.1207/S15327027HC1203_01. PMID 10938914